CLINICAL TRIAL: NCT06593301
Title: The Effect of Education Based on Flip-Face Classroom Model on Nursing Senior Students' Self-Efficacy Regarding Blood and Blood Products Transfusion; Randomized Controlled Study
Brief Title: The Effect of Blood and Blood Products Transfusion Training Based on the Flipped Classroom Model on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: G.Atak
Record Dates: First submitted 2024-07-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Self-efficacy
Keywords: Blood transfusion; flipped classroom; , student

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical learning group (Active Comparator): PRELIMINARY Introductory Information Form, Secure Blood And Blood Products Transfusion Self-Efficacy Scale, Skill Observation Form Routine Applications
  . Theoretical Education; Face in the Classroom Face to Face Training (PPt presentation, verbal lecture, question and answer, discussion, case study etc.)
  Interventions: Other: Flipped classroom model Blood and Gore Based on FCM Products Transfusion Training
- Flipped classroom model group (Experimental): PRELIMINARY Introductory Information Form, Secure Blood And Blood Products Transfusion Self-Efficacy Scale, Skill Observation Form
  Interventions: Other: Flipped classroom model Blood and Gore Based on FCM Products Transfusion Training

INTERVENTIONS:
Other: Flipped classroom model Blood and Gore Based on FCM Products Transfusion Training — Distance Learning; study papers, flowcharts, clinical guides, voiced ppt presentations, skill videos etc. (10 days after face-to-face training before) Theoretical Training Based on FCM; Face to Face In-Class Education (student-centered learning activities, group work, case study, discussion, question answer, etc.)

SUMMARY:
Blood is a living tissue with many vital functions that provide perfusion of organs. Therefore, blood transfusion is a tissue transplant and a complicated treatment method that is applied very frequently. Many reactions may develop during transfusion due to application errors. In this direction, it is necessary to increase the knowledge and skills of nursing students regarding safe blood transfusion during their undergraduate education. On the other hand, self-efficacy is a more comprehensive concept that includes the concepts of knowledge and skills, and self-efficacy perception is considered important in terms of indicating a level of professional development. It is important to use effective teaching methods to increase the knowledge and skills of students and to support their self-efficacy. The flipped classroom model is a teaching method that has the potential to change teaching and learning for nursing education. In the light of this information, this study was planned to determine the effect of education based on the flipped classroom model on the self-efficacy of senior nursing students regarding blood and blood product transfusion.

DETAILED DESCRIPTION:
The study is a non-drug clinical randomized controlled trial and was conducted between February and June 2024. The universe of the study consisted of senior nursing students of the faculty where the study was conducted. In terms of reliability of the study, control group data will be collected first. Criteria for inclusion in the study; Being a senior nursing student and being a volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Being a senior nursing student
* Nursing students who volunteered to participate in the study

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy level | two weeks
  Before the training, data will be collected with the Safe Blood and Blood Products The minimum score that can be obtained from the total scale is 49 and the maximum score is 245. Self-Efficacy Scale and Skill Observation Form (pre-test).
  After the training, students will be evaluated with the Safe Blood and Blood Products Transfusion Self-Efficacy Scale and Skill Observation Form (posttest).The scores that can be obtained from the skill observation form range from 1-30 to 90 and will be evaluated based on the arithmetic average.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH ATAK, Nursing, Principal Investigator — Maltepe,İstanbul,TÜRKİYE, 34854
Locations (1):
- Marmara University Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)